CLINICAL TRIAL: NCT01345903
Title: A Pilot Feasibility and Safety Study Using Robotic Assisted Surgery in Patients With Spine Tumors
Brief Title: Robotic-Assisted Surgery in Treating Patients With Spine Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol needs to be re-designed.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09202; NCI-2011-00691 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Adult Spinal Cord Neoplasm; Spinal Bone Metastases; Spinal Cord Metastases
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (surgery) (Experimental): Patients undergo robotic-assisted surgery using the da Vinci robot
  Interventions: Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo robotic-assisted surgery

SUMMARY:
This pilot clinical trial studies robotic-assisted surgery in treating patients with spine tumors. Robotic-assisted surgery is a less invasive type of surgery for spine tumors and may have fewer side effects and improve recovery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform a small pilot study that will demonstrate the feasibility of neurosurgical spinal procedures using the da Vinci surgical robot.

SECONDARY OBJECTIVES:

I. To compare complication rates, operative time and estimated blood loss with historical controls.

II. To observe wound healing, cerebrospinal fluid (CSF) leaks, neurological injury and hardware failure.

II. Routine imaging of the spinal segment.

OUTLINE:

Patients undergo robotic-assisted surgery using the da Vinci robot.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient has primary or secondary spine tumor based on computed tomography (CT) or magnetic resonance imaging (MRI)
* Karnofsky performance status (PS) of >= 80 or Eastern Cooperative Oncology Group (ECOG) PS 0-1
* Expected survival greater than 3 months
* Patient must be able to understand and sign a study-specific informed consent form

Exclusion Criteria:

* Previous surgery at that specific segment
* Radiation at that specific spinal segment within the last 2 months
* Karnofsky PS < 80 or ECOG PS > 1
* Pregnancy (due to risk of anesthesia)
* The presence of medical conditions which contraindicate general anesthesia
* Unexplained fever or untreated, active infection
* Inability to obtain exposure to allow performance of the planned spine surgical procedure
* History of psychiatric condition or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Complication rates with 95% confidence bounds of +/- 31% or smaller | For 100 days post-surgery
Estimated blood loss | For 100 days post-surgery
Operation duration | At the completion of surgery
Complication rate | For 100 days post-surgery
Demographic and clinical data such as stage, grade and histology | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mike Chen, MD, PhD, Principal Investigator — City of Hope Medical Center